CLINICAL TRIAL: NCT00933010
Title: Osservatorio Regionale Sulla Sindrome metabolicA
Brief Title: Metabolic Syndrome Observation on a Regional Basis
Acronym: ORSA Umbria
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca
Other Study IDs: NIS-CIT-DUM-2008/1
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; lipids; waist circumference; HDL; hypertension
MeSH Terms: conditions — Metabolic Syndrome; Hypertension

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to assess the prevalence of Metabolic Syndrome in Italy on a regional basis, defined according to NCEP/ATPIII Guidelines criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 18 and 75 years
* Signed Informed consent
* Laboratory analysis (lipidic profile and glycemia) performed in the last year

Exclusion Criteria:

* Pregnancy or breast feeding
* Patients enrolled in clinical studies which the aim is to evaluate the efficacy and/or tolerability of anti-hypertensive and/or lipid lowering drugs
* Subjects with serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's successful participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of Metabolic Syndrome in Primary Care Population | July 2009 - March 2010
Concomitant presence of other CV risk factors | July 2009 - March 2010

CONTACTS AND LOCATIONS:
Overall Officials: Mario Mangrella, Study Chair — AstraZeneca S.p.A., R&D; Raffaele Sabia, Study Director — AstraZeneca S.p.A., R&D
Locations (3):
- Italy (3):
  - Research, Foligno
  - Research Site, Perugia
  - Research Site, Terni